CLINICAL TRIAL: NCT00865358
Title: Yoga for Chronic Low Back Pain in a Predominantly Minority Population: A Pilot Randomized Controlled Trial
Brief Title: Yoga for Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT002915
Record Dates: First submitted 2009-02-27; First posted 2009-03-19 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Low Back Pain
Keywords: yoga; complementary alternative medicine; low back pain; minority health; health care disparities; community health centers
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga Group (Experimental): A standardized hatha yoga protocol delivered in 12 weekly classes.
  Interventions: Behavioral: Yoga Group
- Usual care (No Intervention): Participants continue to receive their usual medical care for their back pain

INTERVENTIONS:
Behavioral: Yoga Group — Reproducible standardized 12 week series of hatha yoga classes specifically developed for patients with chronic low back pain and little or no experience with yoga
  Other Names: Hatha yoga classes
  Arms: Yoga Group

SUMMARY:
Chronic low back pain is the most common cause of pain in the United States. Common treatments such as medication, physical therapy, and surgery often do not provide adequate relief. Yoga has shown promise for improving low back pain in studies of predominantly middle class white individuals. We will assess the feasibility and collect preliminary data on yoga for chronic low back pain in predominantly minority individuals in a community health center setting in a low income neighborhood of Boston, Massachusetts. We hypothesize that offering yoga for this population is feasible and will show promising efficacy and safety data.

DETAILED DESCRIPTION:
Promising therapies for chronic low back pain such as yoga need to be studied because conventional treatments such as medication, physical therapy, and surgery frequently do not provide lasting relief. We will use a standardized yoga protocol, developed specifically for this trial by a consensus panel of yoga experts, in a pilot randomized controlled trial for subjects with chronic low back pain. We will recruit 30 predominantly English-speaking minority adults from Boston Medical Center (BMC) and its affiliated clinics with low back pain lasting >12 weeks and an average pain level in the previous week of 4 or more on a scale of 0 to 10 (0 = no pain, 10 = worst possible pain). Subjects will be randomized to a yoga class once per week for 12 weeks (Group 1) or a wait-list control group (Group 2). All subjects will receive their usual medical care and an educational booklet designed for low back pain patients. Primary outcomes are 12 week pain intensity and functional status measured by the Roland Morris Disability scale. Secondary outcomes include analgesic use, health-related quality of life (SF-36), global improvement, subject satisfaction, adverse events, compliance, work status, and health expenditures. Group 2 will be offered yoga classes at 26 weeks. To refine estimates of effect size and further confirm safety of the protocol, we will also collect data from Group 2 during their yoga classes. This pilot will provide preliminary feasibility and efficacy data to plan a future adequately powered randomized controlled trial of yoga for chronic low back pain in predominantly minority subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 18-64 years old. The rationale for including adults only less than 65 years old is that the causes of low back pain in older persons are more likely to be multifactorial (e.g., degenerative disk disease, spinal canal stenosis, fractures) and less likely to be the non-specific muscular type that our yoga protocol was designed to address. A study of yoga for low back pain in individuals > 65 years old is important. However, the ideal design would likely benefit from a yoga protocol specifically designed for this purpose.
2. Current non-specific low back pain lasting at least 12 weeks. Non-specific refers to predominantly muscular and ligamentous causes for the low back pain, and the absence of clear symptoms and signs of other causes of low back pain (e.g., herniated disk). This will be ascertained during the eligibility screening process using the Eligibility Screening Instrument (see Sect. S). This instrument was adapted from eligibility screening tools used in multiple published trials of CAM therapies for chronic low back pain by Karen Sherman PhD and Daniel Cherkin PhD. The instrument uses subject self-report to exclude specific causes of chronic low back pain that are exclusion criteria for the study.
3. Average pain intensity during the week prior to enrollment is 4 or greater on a 0 to 10 numerical pain scale (0=no pain, 10=worst possible pain).
4. Compliant with filling out a 2 week daily pain score dairy during the eligibility screening processes.
5. Ability to comprehend, read, and write English at a level necessary to understand the yoga class instructions and complete data collection forms. Given that this is the first pilot for the yoga protocol and the first trial of yoga for low back pain for predominantly minority adults at BMC and affiliated clinics, we have decided to enhance feasibility by focusing on English speakers first. Our goal is ultimately to study and offer this intervention in other languages commonly spoken by BMC patients (e.g., Spanish). We fully anticipate that this trial will provide the necessary experience to return to the IRB in the near future with a proposal for a pilot trial of Spanish speakers with chronic low back pain.
6. Individuals with sufficient English language ability from all ethnic groups can enroll. However, since this pilot study is specifically targeting minorities with chronic low back pain, we will purposefully allocate 80% (24 of 30) of the openings in the study to minority subjects (ascertained by self-report).
7. Consent to participate.

Exclusion Criteria:

1. Age > 64 years old.
2. Yoga use in the previous 12 months.
3. Inability to understand English at a level necessary to follow yoga class instructions.
4. Pregnancy - although back pain in pregnancy is common and may be amenable to yoga, the causes of the pain are likely different than non specific chronic low back pain in nonpregnant adults.
5. Change in pain medications four weeks or fewer prior to enrollment.
6. Other back pain treatments (e.g., physical therapy, epidural steroid injection, chiropractic, acupuncture) anticipated to begin in the next 6 months or initiated less than four weeks prior to enrollment.
7. Ongoing or planned litigation related to back pain. Ongoing or planned workers' compensation, disability, or personal injury claims related to back pain. Litigation or claims that have been resolved or settled are not exclusion criteria.
8. Back pain by self-report due to specific non-muscular pathologies (e.g., infection, malignancy, fracture); severe or progressive neurological deficits; active substance or alcohol abuse; serious underlying systemic or co-morbid disease that precludes physical or cognitive ability to perform the yoga protocol (see Inclusion Criteria #2 above).
9. Suicidal thoughts detected through the eligibility interview. Those who report suicidal thoughts will immediately be referred to their PCP and/or the BMC Department of Psychiatry.
10. Lack of consent to participate.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-02; Primary Completion 2007-07 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Previous 7 days
Back related function (Modified Roland Morris Disability Scale) | previous 7 days

SECONDARY OUTCOMES:
Pain medication use | previous 7 days
Global improvement | previous 12 weeks
Health Related Quality of Life (SF-36) | previous 7 days
Adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Saper, MD MPH, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Dorchester Multi-Service Center, Dorchester, Massachusetts
  - Codman Square Health Center, Dorchester, Massachusetts